CLINICAL TRIAL: NCT02711189
Title: Oxytocin in Alcohol Use Disorder: A Novel and Translational Approach
Brief Title: Oxytocin in Alcohol Use Disorder
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 160082; 16-AA-0082
Record Dates: First submitted 2016-03-16; First posted 2016-03-17 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-02-22

CONDITIONS: Alcoholism
Keywords: Addiction; Oxytocin; Functional Magnetic Resonance Imaging (fMRI); Alcohol; Cue Reactivity
MeSH Terms: conditions — Alcoholism; Behavior, Addictive | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes

ARMS (2):
- Oxytocin (Active Comparator): Intranasal oxytocin will be delivered on twice daily basis in this crossover trial.
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Within Subject Design
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Oxytocin — Oxytocin nasal spray given in dose 80
  Arms: Oxytocin
Other: Placebo
  Arms: Placebo

SUMMARY:
Background:

Oxytocin is a naturally occurring substance in the body. Studies show that oxytocin may affect how the body responds to alcohol. Researchers believe oxytocin may be a possible treatment for alcoholism.

Objective:

To test whether the hormone oxytocin affects the brain reward system. To see if it affects how people respond to alcohol and other rewarding things in life like food and seeing loved ones.

Eligibility:

Men ages 21-55 who have an alcohol use disorder.

Design:

Participants will have two 6-day inpatient study visits. They will have:

* Study medication or placebo given twice daily as a nasal spray.
* Height and weight measured.
* Medical history.
* Blood and urine tests.
* Breath tested for alcohol.
* Electrocardiogram.
* An alcohol administration session. In a bar-like room, where participants will consume four alcoholic drinks.
* Magnetic resonance imaging (MRI). The MRI scanner is a metal cylinder in a strong magnetic field. Participants will lie on a table that slides in and out of the cylinder. A device called a coil will be placed over their head. Participants will complete tasks on a computer screen.
* In another alcohol session. they will drink an alcoholic beverage then answer questions. Participants will get a tab for eight more drinks ($3.00 per drink). They may drink any of the drinks or take the money. Participants will hold and smell a glass of water and their favorite alcoholic drink.
* Heart rate and blood pressure will be monitored.
* Saliva samples will be collected
* Computer tasks and questionnaires.

About one week after the end of visit 2, participants will return to clinic for a follow-up visit. Symptoms and side effects will be evaluated.

DETAILED DESCRIPTION:
Objective:

There is compelling evidence to support that the neuropharmacology of oxytocin (OT) warrants further investigation as a potential therapeutic agent for addiction. To that end, the link between OT and dopaminergic pathways, with respect to motivated behaviors such as drug and social reward, is important to establish as a mechanism. Although preliminary clinical findings suggest a role of OT to treat withdrawal in alcoholic individuals, there is no direct human evidence on the effects of OT administration on dopamine release. Additionally, there is no direct human evidence on the effects of OT on the subjective response to alcohol. There have been no studies investigating the differential effect, if any, of OT, on the neurobehavioral response to various rewarding stimuli including alcohol, food and social reward. We propose, therefore, to investigate whether intranasal administration of OT is able to significantly reduce subjective response to alcohol, alcohol cue-induced craving and self-administration, as well as to examine the neural response to social, alcohol and food stimuli.

Study Population:

32 (24 completers) males with Alcohol Use Disorder (AUD) as defined by DSM-5 and non-treatment seekers for AUD.

Design:

A within-subject, double-blind placebo-controlled study investigating the effect of intranasal OT on the response to alcohol challenge, cue reactivity and alcohol self-administration, and the neural response to rewarding stimuli. Outcome measures: a) effect of OT on subjective response to cumulative alcohol challenge, cue reactivity and alcohol self-administration; b) neurobehavioral response to social, alcohol and food stimuli.

Outcome measures:

A) effect of OT on subjective response to cumulative alcohol challenge, cue reactivity and alcohol self-administration; B) neurobehavioral response to social, alcohol and food stimuli.

ELIGIBILITY:
* INCLUSION CRITERIA:
* 21-55 year old male subjects. Justification: women will not be included due to: 1) the confound of the estrogen-modulating effect of OT; 2) the need to control for menstrual cycle phase across repeated days of study procedures which would significantly limit the feasibility of the study
* Must meet DSM-5 criteria for AUD based on the SCID
* Right handed

EXCLUSION CRITERIA:

* Non-drinkers (alcohol-naive individuals or current abstainers).
* Currently seeking treatment to reduce or stop alcohol use.
* Current diagnosis of substance use disorder other than nicotine as determined by DSM-5.
* Current clinically significant major depression or anxiety; or lifetime diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, or obsessive compulsive disorder.
* Lifetime history of suicide attempts.
* Contraindications for MRI scanning, including metal in body that are contraindicated for MRI (such as implants, pacemaker, prostheses, shrapnel, irremovable piercings), left-handedness, claustrophobia or unable to lie comfortably supine for up to 2 hours in the and MRI scanner as determined from history and physician examination and the MRI safety form.
* BMI>40 or if Investigators determine that subject s body shape precludes acquisition of an adequate MRI scan.
* Unable to provide a negative urine drug test (UDT).
* Medical contraindications: Current clinically significant disease, including CNS, seizures, cardiovascular, hypertension, arrhythmias, glaucoma, respiratory, gastrointestinal, hepatic, renal, endocrine, or reproductive disorders as determined by history and clinical exam at screening. Specifically, unstable hypertension, clinically significant EKG abnormalities, GFR rate > 60ml/min, liver cirrhosis, AST or ALT > 3X the upper normal limit, hemoglobin < 10.5 g/dl.
* Participants who have significant alcohol withdrawal symptoms as defined by CIWA-Ar>8.
* History of alcohol related seizures
* Requirement for or use in the past two weeks of psychoactive medications (four weeks for fluoxetine).
* Use of prescription or OTC medications known to interact with alcohol within 2 weeks of the study. These include, but may not be limited to: isosorbide, nitroglycerine, benzodiazepines, warfarin, anti-depressants such as amitriptyline, clomipramine and nefazodone, anti-diabetes medications such as glyburide, metformin and tolbutamide, H2-antagonists for heartburn such as cimetidine and ranitidine, muscle relaxants, anti-epileptics including phenytoin and phenobarbital codeine, and narcotics including darvocet, percocet and hydrocodone. Drugs known to inhibit or induce enzymes that metabolize alcohol should not be used for 4 weeks prior to the study. These include chlorzoxazone, isoniazid, metronidazole and disulfiram. Cough-and-cold preparations, which contain anti-histamines, pain medicines and anti-inflammatories such as aspirin, ibuprofen, acetaminophen, celecoxib and naproxen, should be withheld for at least 72 hours prior to each study session.
* History of hypersensitivity to oxytocin.
* Clinically significant electrolyte abnormalities, current rhinitis or use of vasoconstricting medications or prostaglandins
* Head trauma with loss of consciousness for more than 30 minutes.
* Any individuals with colorblindness that would prevent them from completing the Stroop task.
* Any other reason for which the Investigators will determine that it is not in the best interest of the participant to take part in this research.

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03-08; Primary Completion 2019-02-22 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Alcohol Craving, Self-Administration | Ongoing
Stimulation Sedation; Cognitive Performance | Ongoing
BOLD response cognitive tasks and cues | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Mary R Lee, M.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)

REFERENCES:
- [Background] Pedersen CA, Smedley KL, Leserman J, Jarskog LF, Rau SW, Kampov-Polevoi A, Casey RL, Fender T, Garbutt JC. Intranasal oxytocin blocks alcohol withdrawal in human subjects. Alcohol Clin Exp Res. 2013 Mar;37(3):484-9. doi: 10.1111/j.1530-0277.2012.01958.x. Epub 2012 Oct 1. PMID 23025690
- [Background] McGregor IS, Bowen MT. Breaking the loop: oxytocin as a potential treatment for drug addiction. Horm Behav. 2012 Mar;61(3):331-9. doi: 10.1016/j.yhbeh.2011.12.001. Epub 2011 Dec 14. PMID 22198308